CLINICAL TRIAL: NCT02305771
Title: Contributions From the Analysis of Graphs for Identification of Neural Cliques
Acronym: BRAINGRAPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-A01461-46; 35RC14_9849_BRAINGRAPH (Other: Rennes University Hospital)
Record Dates: First submitted 2014-11-28; First posted 2014-12-03 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Healthy volunteers (Other): 20 healthy volunteers will undergo an inclusion visit in order to check inclusion and non inclusion criteria.
  Then will be performed:
  * Electroencephalography
  * MRI
  Interventions: Device: Electroencephalography; Device: MRI

INTERVENTIONS:
Device: Electroencephalography
Device: MRI

SUMMARY:
The aim of the study is to demonstrate that our semantic knowledge (elements of our long-term memory and the process we use them) respond to a graphic organisation and gather together following accurate patterns called cliques (neural networks).

DETAILED DESCRIPTION:
Electroencephalography (EEG) with very High spatial Resolution (HR) (EEG-HR, 256 electrodes) allows for a better understanding of the global and local activity of the cerebral neocortex.

In 2012, following publications by Claude Berrou and Vincent Gripon's Internet, introducing new principles of coding information based on graphical representations in connectionist networks, we approached this team to test biological plausibility of this theory in vivo with EEG.

The central concept is the mental information, defined as all elements of knowledge acquired by the long-term memory on which the reason can build to try to respond to new problems. According to this new theory, these elements of knowledge called qualia or features should be connected within cliques networks. However, we currently do not have graphs comparing methods to measure a good index of both spatial and topological similarity between graphs with high resolution electroencephalography.

For this new study, we propose to combine the strengths of several existing methods of graph comparison which, on top of this, will be especially adapted to the specific context of the analysis of the graphs in the cerebral cortex.

The skills used are diverse: information theory, mathematics, graph theory, computer science, neuropsychology, signal processing and neurology.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Right-handed ;
* French native speaker
* Having given written informed consent

Exclusion Criteria:

* Presence of any psychiatric, neuropsychological and developmental disorder
* Any uncorrected visual impairment
* Any trouble or delay in learning to read / speak french
* Fully bilingual or multilingual
* Medication, treatment and / or substances that may alter or modify brain functions
* Pregnancy, breast feeding
* Persons under major legal protection and/or deprived of liberty

MRI-related criterions

* Cardiac pacemaker or implanted defibrillator
* Iron-magnetic surgical clips
* Cochlear implant
* Intra-ocular or brain foreign bodies
* Less than 4 weeks-old stents, less than 6 weeks-old osteosynthesis materials
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2015-11-20 (Actual); Study Completion 2015-11-20 (Actual)

PRIMARY OUTCOMES:
Three main criteria are to be considered to validate the tool for measuring the similarity between the graphs obtained | 2 years
  Despite the intra-individual variability, the same object or the same sound repeated several times should generate the most similar connectivity graphs Despite the inter-individual variability, analysis of connectivity graphs must also report high similarity indices between individuals on the same stimuli or stimuli sharing the same semantic properties even if subjects are different.
  At the stage of conceptual analysis of stimuli, or from 175 ms after the presentation of the image or sound, the analysis of connectivity graphs should reveal strong similarity indices for several different images of the same object (independence to the visual representation); for picture and sound representing the same object (independence to the sensory modality) or two objects belonging to the same semantic category (conceptual similarity, eg: orange, lemon). Indeed, these objects share common characteristics / semantic dimensions (eg mobile vs. stationary or living vs. non-living etc.).
Estimate the plausibility of the results obtained with our method directly from the graphs | 2 years
  The density (ie: the ratio between the number of links in a given graph on the total possible number of links), the diameter (ie: the longest path in a graph), the average degree (ie: the average number of links connected to each node), the clustering (ie: the density of connections to a group of nodes with the rest of the network) and other parameters will be compared in terms of standard values available in the literature but also with tools that help to calculate the semantic distance between words such as WordNet and many others.

SECONDARY OUTCOMES:
Judgement of the quality of the measurement on simulated data in the laboratory test our method for measuring the similarity between the graphs | 2 years
  A computer model of neural network populations in which the experimenter knows in advance where the sources are allows him to test the reliability of his methods while reconstructing graphs and judging their similarity. [8] Finally, the quality of the results about the identification of neural cliques (or complete graphs) could be compared to the artificial neural network model we develop elsewhere [1, 9 and 10]. This model indicates that the distribution of neural cliques (in response to density and efficiency problems) follows a simple principle that we should find in the brain. For example, it is reasonable to think there are many cliques (or complete graphs) at the scale of a small brain region while those cliques are rare when considering spatially distant sources. It is an organization called "small-worlds" and which is classical for the neural networks in the cerebral cortex

CONTACTS AND LOCATIONS:
Locations (1):
- Rennes University Hospital, Rennes, France

REFERENCES:
- [Result] Mheich A, Dufor O, Yassine S, Kabbara A, Biraben A, Wendling F, Hassan M. HD-EEG for tracking sub-second brain dynamics during cognitive tasks. Sci Data. 2021 Jan 27;8(1):32. doi: 10.1038/s41597-021-00821-1. PMID 33504796